CLINICAL TRIAL: NCT00626340
Title: Measurement of GABA and Neurosteroid Levels in Women With Menopausal Major Depression Before and After Treatment With Estrogen Alone, Fluoxetine Alone, or Estrogen and Fluoxetine and Normal Controls Before and After Treatment With Estrogen
Brief Title: Brain Imaging Study in Menopausal Women With and Without Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9907010780
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Menopause; Depression
Keywords: menopause; women; major depressive disorder; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MDD diagnosis and Estrogen treatment (Active Comparator): Menopausal women between the ages of 40-70 diagnosed with Major Depressive Disorder receiving treatment with estrogen alone.
  Interventions: Drug: MDD diagnosis and Estrogen treatment
- MDD diagnosis and Fluoxetine treatment (Active Comparator): Menopausal women between the ages of 40-70 diagnosed with Major Depressive Disorder receiving treatment with fluoxetine alone.
  Interventions: Drug: MDD diagnosis and Fluoxetine treatment
- MDD diagnosis with both Estrogen and Fluoxetine treatment (Active Comparator): Menopausal women between the ages of 40-70 diagnosed with Major Depressive Disorder receiving treatment with estrogen and fluoxetine combined.
  Interventions: Drug: MDD diagnosis with both Estrogen and Fluoxetine treatment
- No depression and estrogen treatment (Active Comparator): Non-depressed menopausal women between the ages of 40-70 receiving treatment with estrogen alone.
  Interventions: Drug: No depression and estrogen treatment

INTERVENTIONS:
Drug: MDD diagnosis and Estrogen treatment — Treatment for major depressive disorder occurring in the context of the menopause while participating in brain imaging sessions pre and post treatment. Women receiving treatment for depression will be compared to normal controls receiving estrogen only for physical symptoms of menopause.
  Arms: MDD diagnosis and Estrogen treatment
Drug: MDD diagnosis and Fluoxetine treatment — Menopausal women between the ages of 40-70 diagnosed with Major Depressive Disorder receiving treatment with fluoxetine alone.
  Arms: MDD diagnosis and Fluoxetine treatment
Drug: MDD diagnosis with both Estrogen and Fluoxetine treatment — Menopausal women between the ages of 40-70 diagnosed with Major Depressive Disorder receiving treatment with estrogen and fluoxetine combined.
  Arms: MDD diagnosis with both Estrogen and Fluoxetine treatment
Drug: No depression and estrogen treatment — Control participants with no MDD diagnosis received estrogen only for the treatment of physical symptoms of menopause.
  Arms: No depression and estrogen treatment

SUMMARY:
The purpose this study is to measure cortical gama-aminobutyric acid levels (GABA) levels in menopausal women with major depressive disorder and healthy subjects using nuclear magnetic resonance spectroscopy (MRS). Measurements will be compared in 1) menopausal healthy subjects before and after estrogen replacement, and after fourteen days of medroxyprogesterone administration; and 2) in depressed menopausal subjects before and after treatment of their depression with antidepressant alone, estrogen alone or antidepressant plus estrogen. Cortical GABA levels will be correlated with plasma GABA and neurosteroid levels. Neurosteroids to be measured include progesterone, allopregnanolone, pregnenolone, and pregnenolone sulfate.

ELIGIBILITY:
Inclusion criteria for Depressed Patients:

* Aged 40-70 years and able to give voluntary written informed consent.
* Meet DSM-IV criteria for major depression based on a structured clinical interview (SCID).
* Have no medical contraindication to estrogen. (This will include written documentation of a recent normal gynecological evaluation and mammogram).
* A minimum score of 25 on the 25-item Hamilton Depression Rating Scale on initial baseline rating which does not show improvement during the one-week observation period.
* Perimenopausal subjects will be those who have had irregular menses of either <21 days or >35 days for the previous six months to one year. Postmenopausal subjects will be those with no menstrual cycles and no hormone therapy for at least one year and serum FSH >45.

Exclusion criteria:

* Meeting DSM-IV for any other Axis I disorder.
* A history of serious medical or neurological illness, including (but not limited to) major cardiovascular disease, severe hypertension, intracranial mass lesions, seizure disorder, severe hepatic or renal disease, unstable endocrine or metabolic disease, and unstable hematologic disease.
* A history of moderate to severe endometriosis; milder cases will require subject's Gynecologists permission to participate.
* Use of anticonvulsants or benzodiazepines within the last month.
* Use of psychotropic medication in last week (except as stated above).
* Use of alcohol within last month.
* Current pregnancy (for the perimenopausal subjects).
* Positive urine drug screen.
* Metallic implants.

Inclusion Criteria for Healthy Subjects:

* No DSM-IV psychiatric or substance abuse diagnosis by structured diagnostic interview (SCID).
* No medical contraindication to estrogen (this will include written documentation of a recent normal gynecological exam with mammogram).
* Matched to depressed patients by age and menopausal status.
* Have no menstrual cycles or hormone therapy for at least one year or irregular menses of either <21 days or 35 days for the previous six months to one year.

Exclusion Criteria for Healthy Subjects:

* Medical, neurologic or cerebrovascular disorder (CVA, seizure disorder, etc.).
* Evidence of substance use on urine toxicology screen done upon recruitment.
* Current treatment with psychoactive medication.
* Diabetes controlled by means other than diet.
* Use of alcohol within last month.
* Implanted metallic devices.
* Positive urine drug screen.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1999-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, MD, Principal Investigator — University of Pennsylvania School of Medicine Department of Psychiatry
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Weissman MM, Klerman GL. Sex differences and the epidemiology of depression. Arch Gen Psychiatry. 1977 Jan;34(1):98-111. doi: 10.1001/archpsyc.1977.01770130100011. PMID 319772
- [Background] Steiner M. Female-specific mood disorders. Clin Obstet Gynecol. 1992 Sep;35(3):599-611. doi: 10.1097/00003081-199209000-00020. PMID 1521388
- [Background] Pariser SF. Women and mood disorders. Menarche to menopause. Ann Clin Psychiatry. 1993 Dec;5(4):249-54. doi: 10.3109/10401239309148824. PMID 8312982
- [Background] Pearlstein TB. Hormones and depression: what are the facts about premenstrual syndrome, menopause, and hormone replacement therapy? Am J Obstet Gynecol. 1995 Aug;173(2):646-53. doi: 10.1016/0002-9378(95)90297-x. PMID 7645647
- [Background] Nicol-Smith L. Causality, menopause, and depression: a critical review of the literature. BMJ. 1996 Nov 16;313(7067):1229-32. doi: 10.1136/bmj.313.7067.1229. PMID 8939110
- [Background] Schmidt PJ, Rubinow DR. Menopause-related affective disorders: a justification for further study. Am J Psychiatry. 1991 Jul;148(7):844-52. doi: 10.1176/ajp.148.7.844. PMID 2053622
- [Background] Arpels JC. The female brain hypoestrogenic continuum from the premenstrual syndrome to menopause. A hypothesis and review of supporting data. J Reprod Med. 1996 Sep;41(9):633-9. PMID 8887186
- [Background] Lopez-Jaramillo P, Teran E, Molina G, Rivera J, Lozano A. Oestrogens and depression. Lancet. 1996 Jul 13;348(9020):135-6. doi: 10.1016/s0140-6736(05)64656-9. No abstract available. PMID 8676707
- [Background] Ditkoff EC, Crary WG, Cristo M, Lobo RA. Estrogen improves psychological function in asymptomatic postmenopausal women. Obstet Gynecol. 1991 Dec;78(6):991-5. PMID 1658700
- [Background] Schneider MA, Brotherton PL, Hailes J. The effect of exogenous oestrogens on depression in menopausal women. Med J Aust. 1977 Jul 30;2(5):162-3. doi: 10.5694/j.1326-5377.1977.tb99116.x. PMID 197385
- [Background] Thomson J, Oswald I. Effect of oestrogen on the sleep, mood, and anxiety of menopausal women. Br Med J. 1977 Nov 19;2(6098):1317-9. doi: 10.1136/bmj.2.6098.1317. PMID 338104
- [Background] Berlanga C. Potentiating effect of estrogen in a patient with treatment-resistant depression. J Clin Psychiatry. 1988 Dec;49(12):504. No abstract available. PMID 2848799
- [Background] Oppenheim G. A case of rapid mood cycling with estrogen: implications for therapy. J Clin Psychiatry. 1984 Jan;45(1):34-5. PMID 6141158
- [Background] Freeman EW, Purdy RH, Coutifaris C, Rickels K, Paul SM. Anxiolytic metabolites of progesterone: correlation with mood and performance measures following oral progesterone administration to healthy female volunteers. Neuroendocrinology. 1993 Oct;58(4):478-84. doi: 10.1159/000126579. PMID 7904330
- [Background] Halbreich U, Petty F, Yonkers K, Kramer GL, Rush AJ, Bibi KW. Low plasma gamma-aminobutyric acid levels during the late luteal phase of women with premenstrual dysphoric disorder. Am J Psychiatry. 1996 May;153(5):718-20. doi: 10.1176/ajp.153.5.718. PMID 8615423
- [Background] Krystal JH, Karper LP, Seibyl JP, Freeman GK, Delaney R, Bremner JD, Heninger GR, Bowers MB Jr, Charney DS. Subanesthetic effects of the noncompetitive NMDA antagonist, ketamine, in humans. Psychotomimetic, perceptual, cognitive, and neuroendocrine responses. Arch Gen Psychiatry. 1994 Mar;51(3):199-214. doi: 10.1001/archpsyc.1994.03950030035004. PMID 8122957
- [Background] Mazure C, Nelson JC, Price LH. Reliability and validity of the symptoms of major depressive illness. Arch Gen Psychiatry. 1986 May;43(5):451-6. doi: 10.1001/archpsyc.1986.01800050053006. PMID 3964024
- [Background] Petty F, Kramer GL, Gullion CM, Rush AJ. Low plasma gamma-aminobutyric acid levels in male patients with depression. Biol Psychiatry. 1992 Aug 15;32(4):354-63. doi: 10.1016/0006-3223(92)90039-3. PMID 1420649
- [Background] Rothman DL, Petroff OA, Behar KL, Mattson RH. Localized 1H NMR measurements of gamma-aminobutyric acid in human brain in vivo. Proc Natl Acad Sci U S A. 1993 Jun 15;90(12):5662-6. doi: 10.1073/pnas.90.12.5662. PMID 8516315
- [Background] Squires RF, Saederup E. Antidepressants and metabolites that block GABAA receptors coupled to 35S-t-butylbicyclophosphorothionate binding sites in rat brain. Brain Res. 1988 Feb 16;441(1-2):15-22. doi: 10.1016/0006-8993(88)91378-9. PMID 2833998
- [Background] Wisner KL, Wheeler SB. Prevention of recurrent postpartum major depression. Hosp Community Psychiatry. 1994 Dec;45(12):1191-6. doi: 10.1176/ps.45.12.1191. PMID 7868100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at an outpatient research facility located at Yale University in New Haven, CT.
Groups:
- All Participants: This study was conducted at Yale University almost two decades ago. Our group at the University of Pennsylvania only has very basic information about this study. This includes the number of participants, which was 18, and the fact that no adverse events occurred. Staff members at the University of Pennsylvania do not have access to any additional study data. The contact person who initially entered this study protocol information is no longer at the University of Pennsylvania and we are unable to contact for additional information.
Period: Overall Study
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: As far as we know, data was never analyzed for this study. We only know that 18 participants completed.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Continuous [unit: years] — Population: UPenn does not have access to the data collected for this study. We are only using the information entered in the protocol section for very basic details in the results section (i.e, number of participants completed). The original contact person for this protocol is not reachable.
Sex: Female, Male — Population: UPenn does not have access to the data collected for this study. We are only using the information entered in the protocol section for very basic details in the results section (i.e, number of participants completed). The original contact person for this protocol is not reachable.

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Cortical GABA Levels in 4 Groups of Subjects Using Estrogen Alone, Fluoxetine Alone, Estrogen and Fluoxetine Combined in Pre and Post 4.0T Magnetic Resonance Spectroscopy Sessions.
Description: This study was conducted at Yale University almost two decades ago. Our group at the University of Pennsylvania only has very basic information about this study. This includes the number of participants, which was 18, and the fact that no adverse events occurred. Staff members at the University of Pennsylvania do not have access to any additional study data. The contact person who initially entered this study protocol information is no longer at the University of Pennsylvania and we are unable to contact for additional information.
  We only know that 18 participants completed, but as far as we know data was never analyzed for these 18 participants.
Time Frame: Healthy controls will undergo scans pre and post 3 weeks of estrogen treatment. Women with depression will undergo scans pre and post 6 weeks of treatment with estrogen alone, estrogen and fluoxetine, or fluoxetine alone
Population: UPenn does not have access to the data collected for this study. We are only using the information entered in the protocol section for very basic details in the results section (i.e, number of participants completed). The original contact person for this protocol is not reachable.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Time Frame: Entire study duration
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No